CLINICAL TRIAL: NCT06913751
Title: Impact of Air Quality on the Effectiveness of Standard of Care Therapy in Children With Autism Spectrum Disorder: A Prospective Longitudinal Study
Status: Not yet recruiting | Type: Observational
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Sheffali Gulati, Professor, All India Institute of Medical Sciences
Other Study IDs: AIIMSA2566
Record Dates: First submitted 2025-03-31; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Autism Spectrum Disorder
Keywords: autism spectrum disorder; Air pollution
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Three millilitres of blood sample will be collected from every 5th patient from each group, at the end of 6 months follow up,. Samples will be collected only from those patients who provide consent for the same. A total of 10 samples, 5 from each group will be collected and analysed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Children with autism spectrum disorder followed up during the months with lower air pollution: * First group of children with autism spectrum disorder who meet the inclusion and exclusion criteria will be enrolled in the study after due informed consent in the month of April 2025.
  * The children will be followed up for a period of 6 months till September 2025 when they will be evaluated for primary outcome- CARS-2 score and other secondary outcomes-behavioural issues/sleep issues/cognitive ability.
  * They will further be followed up for the next 6 months till March 2026 to be evaluated for secondary outcomes.
  Interventions: Behavioral: standard of care
- Children with autism spectrum disorder followed up during the months with higher air pollution: * Second group of children with autism spectrum disorder who meet the inclusion and exclusion criteria will be enrolled in the study after due informed consent in the month of October 2025.
  * The children will be followed up for a period of 6 months till March 2026 when they will be evaluated for primary outcome- CARS-2 score and other secondary outcomes-behavioural issues/sleep issues/cognitive ability.
  * They will further be followed up for the next 6 months till September 2026 to be evaluated for secondary outcomes.
  Interventions: Behavioral: standard of care

INTERVENTIONS:
Behavioral: standard of care — standard of care therapy with behavioural and occupational therapy along with other pharmacological therapy as required

SUMMARY:
1. Air quality is a growing concern for health and environment and is one of the modifiable environmental factors. There is growing evidence that a complex interplay of genetic and epigenetic factors like environmental factors, underlies the pathophysiology of ASD. Behavioural issues, sleep habits and cognitive abilities play a significant role in the quality of life of both the affected children and their caregivers
2. Few studies have shown that there is an increased incidence of ASD in children born to mothers exposed to higher levels of air pollution in pregnancy. However, no studies on the effect of air quality on the severity of autism. There are limited studies on the association of air pollution with childhood behaviour and cognitive abilities, especially in neurodevelopmental disorders. No evidence on the impact of air quality on the effectiveness of therapy/standard of care in children with autism, as well as on their sleep habits and behaviour.

Our study aims to add to this growing body of evidence of the effect of air pollution on ASD in children.

DETAILED DESCRIPTION:
* All Children with ASD aged 3-12 years attending pediatric neurology OPD and autism clinic will be screened for eligibility.
* Those children fulfilling the inclusion and exclusion criteria will be enrolled into the study.
* First group of children will be enrolled in the month of April 2025 and followed up for a period of 6 months during which the air pollution levels are lower (Average AQI <200) (April to September 2025), following which the primary assessment will be done in the end of September 2025 and then subsequently followed up again for another 6 months. At the end of 1 year, i.e. in the end of March 2026, they will undergo secondary assessment.
* Second group of children will be enrolled in the month of October 2025 and followed up for a period of 6 months during which the air pollution levels are higher (Average AQI >200) (October to March 2026), following which the primary assessment will be done in the end of March 2026 and then subsequently followed up again for another 6 months. At the end of 1 year, i.e. in the end of September 2026, they will undergo secondary assessment.
* Matching of both groups: Both the groups will be matched for all possible confounders

  1. Age
  2. Gender
  3. Socioeconomic status
  4. Household fuel
  5. Severity of autism
  6. Any smoker at home
  7. Cooking method used at home
  8. Overcrowding
  9. Use of AC/Cooler/Fan/Heater as appropriate
  10. BMI
  11. Other relevant clinical and medical details
* Bias: In order to avoid possible observer bias, the baseline assessment will be done and intervention module will be provided by the primary investigator. The follow up assessments at 6 and 12 months will be done by another DM senior resident from the division of child neurology.

Intervention and management of enrolled patients

* Informed consent will be taken from parents/legally acceptable representatives for the study
* Baseline demographic details and following evaluation will be done - Autism severity assessment using CARS -2 score Cognitive assessment using VABS/DP-3/MISIC Behavioural assessment using CBCL questionnaire Screening for sleep related disorders using CSHQ score Group I- Children with autism spectrum disorder followed up during the months with lower air pollution
* First group of children with autism spectrum disorder who meet the inclusion and exclusion criteria will be enrolled in the study after due informed consent in the month of April 2025.
* Their demographic details including place of residence will be collected at baseline.
* The children will also be evaluated for their baseline CARS score, DQ/SQ/IQ, sleep related disorders and behavioural issues using standardised validated tools as described above.
* The children will be followed up for a period of 6 months till September 2025 when they will be evaluated for primary outcome- CARS-2 score and other secondary outcomes-behavioural issues/sleep issues/cognitive ability.
* They will further be followed up for the next 6 months till March 2026 to be evaluated for secondary outcomes.
* At the end of 12 month follow up period, the children will again be evaluated for CARS-2 score, DQ/SQ/IQ, sleep related disorders and behavioural issues using standardised validated tools as described above.
* Data on exposure to air pollution (daily average PM 2.5 and PM 10 levels) will be collected for the total follow up period of 1 year based on the nearest air pollution monitoring site of CPCB.
* Those children identified with sleep issues in the CSHQ questionnaire will be managed as per the standard guidelines and will undergo actigraphy and polysomnography as and when warranted.
* In children with behaviour issues, standard of care will be provided in the form of anti-psychotic medications and other behavioural interventions.

Group II- Children with autism spectrum disorder followed up during the months with higher air pollution

* Second group of children with autism spectrum disorder who meet the inclusion and exclusion criteria will be enrolled in the study after due informed consent in the month of October 2025.
* Their demographic details including place of residence will be collected at baseline.
* The children will also be evaluated for their baseline CARS score, DQ/SQ/IQ, sleep related disorders and behavioural issues using standardised validated tools as described above.
* The children will be followed up for a period of 6 months till March 2026 when they will be evaluated for primary outcome- CARS-2 score and other secondary outcomes-behavioural issues/sleep issues/cognitive ability.
* They will further be followed up for the next 6 months till September 2026 to be evaluated for secondary outcomes.
* At the end of 12 month follow up period, the children will again be evaluated for CARS-2 score, DQ/SQ/IQ, sleep related disorders and behavioural issues using standardised validated tools as described above.
* Data on exposure to air pollution(daily average PM 2.5 and PM 10 levels)will be collected for the total follow up period of 1 year based on the nearest air pollution monitoring site of CPCB.
* Those children identified with sleep issues in the CSHQ questionnaire will be managed as per the standard guidelines and will undergo actigraphy and polysomnography as and when warranted.
* In children with behaviour issues, standard of care will be provided in the form of anti-psychotic medications and other behavioural interventions.

Blood Sample Analysis for Nuclear Chromatin To assess the gene expression changes due to air pollution, epigenetic mark on histone proteins, a core component of chromatin that needs to be closed or open state for transcriptional changes, can be measured. The H3 trimethylated at lysine 4 (H3K4me3) represents an open chromatin state representing active transcription. Chromatin immunoprecipitation using antibody detecting H3K4me3 followed by sequencing of the DNA fragments (ChIP-Seq) will determine active or poised transcription. Hence, the objective of the study is to perform ChIP-Seq analysis from peripheral blood samples to visualize the global change in transcription. Detection of transcriptional change would lead to further study to assess open vs. closed chromatin state. This will be determined by ATAC-Seq that detects chromatin states and subsequent RNA-Seq from same sample that determine RNA expression level as an indicator of transcription.

Three millilitres of blood sample will be collected from every 5th patient from each group, at the end of 6 months follow up, for the above analysis. Samples will be collected only from those patients who provide consent for the same. A total of 10 samples, 5 from each group will be collected and analysed.

Informed consent Eligible children will be enrolled only after receiving written informed consent from parents/guardian. Parents will be explained about the voluntary nature of participation in the study and the option to withdraw from the study at any point in time.

Ethical considerations Parents or LAR of the eligible children will be approached and explained regarding the study. Only those children whose parents/LAR give written informed consent will be enrolled in the study. The study protocol will be submitted to the AIIMS Institute Ethics Committee for approval and the study will be initiated only after such an approval is received.

ELIGIBILITY:
Inclusion Criteria:1. Children aged 3- 12 years diagnosed with ASD according to DSM -V criteria and those who have received standard of care for less than 6 months at the time of screening and enrolment 2. Resident of Delhi-NCR

-

Exclusion Criteria:

1. Other known secondary causes of ASD like Fragile-X Syndrome, Down Syndrome, Tuberous sclerosis, etc.
2. ASD with known metabolic disorders
3. ASD with drug refractory epilepsy

   -

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with ASD based on DSM -V criteria between 3- 12 years of age attending the Pediatric Neurology OPD and Autism clinic, in Department of Pediatrics, at AIIMS, New Delhi
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
To compare the effectiveness of standard of care therapy, in terms of change in CARS score after 6 months follow up, in two groups of children with autism spectrum disorder, during months with high air pollution and low air pollution, based on AQI | 6 months
  Difference in the change in mean CARS score between the two groups at 6 months follow up

SECONDARY OUTCOMES:
To compare the effectiveness of standard of care therapy, in terms of change in CARS score after 12 months follow up, in two groups of children with autism spectrum disorder, during months with high air pollution and low air pollution, based on AQI | 12 months
  Difference in the change in mean CARS score between the two groups at 12 months follow up
To compare the impact on cognitive ability, as measured in terms of change in DQ/SQ/IQ after 6 months follow up, in two groups of children with autism spectrum disorder, during months with high air pollution and low air pollution, based on AQI | 12 months
  Difference in the change in mean DQ/IQ/SQ score between the two groups at 6 and 12 months follow up
To compare the impact on sleep habits, as measured in terms of change in CSHQ score after 6 months follow up, in two groups of children with autism spectrum disorder, during months with high air pollution and low air pollution, based on AQI | 12 months
  Difference in the change in mean CSHQ score between the two groups at 6 and 12 months follow up
To compare the impact on behavioral profile, as measured in terms of change in CBCL score after 6 months follow up, in two groups of children with autism spectrum disorder, during months with high air pollution and low air pollution, based on AQI | 12 months
  Difference in the change in mean CSHQ score between the two groups at 6 and 12 months follow up
To assess the corelation between the air quality parameters (PM2.5, PM10) and the severity of autism spectrum disorder/sleep issues/behavioural issues and cognition at the end of 6 months follow up | 12 months
  Corelation between average PM 2.5, PM 10 levels during the 6 and 12 month follow up period and CARS score/CHSQ score/CBCL score/IQ
To assess for genetic changes by comparing the global change in transcription, between children receiving standard of care during high pollution months and those receiving during low pollution months | 6 months
  To detect transcriptional change, and compare it between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: sheffali gulati, MD, Principal Investigator — All India Institute of Medical Sciences, New Delhi, Delhi 110029

IPD SHARING:
Plan to Share IPD: No